CLINICAL TRIAL: NCT07192848
Title: Efficacy and Safety of Adebrelimab Plus Apatinib in Patients With Advanced Hepatocellular Carcinoma Previously Treated With Systemic Therapy: A Single-arm, Phase II Study
Brief Title: Adebrelimab + Apatinib in Advanced HCC Post-Systemic Therapy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Song Peng (Other)
Responsible Party: Sponsor-Investigator, Song Peng, Principal Investigator, Cancer Hospital Chinese Academy of Medical Science, Shenzhen Center
Organization: Cancer Hospital Chinese Academy of Medical Science, Shenzhen Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YW2025-17-1
Record Dates: First submitted 2025-08-13; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Hepatocellular Carcinoma Non-resectable
Keywords: Adebrelimab; Apatinib; Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adebrelimab + Apatinib Treatment Arm (Experimental): This arm involves patients receiving adebrelimab (1200mg, intravenous infusion on D1, Q3W) combined with apatinib (250mg, oral, QD). Treatment continues until intolerable toxicity, withdrawal of consent, disease progression, or other protocol - defined criteria.
  Interventions: Drug: Adebrelimab + Apatinib

INTERVENTIONS:
Drug: Adebrelimab + Apatinib — Adebrelimab: A fixed dose of 1200 mg is administered as an intravenous infusion over 30 minutes (not less than 20 minutes and not more than 60 minutes, including the flushing phase), once every 3 weeks (Q3W). The interval between two administrations should not be less than 12 days.
  The maximum treatment duration is 6 courses.
  Apatinib: 250 mg, once daily (QD), taken orally within half an hour after a meal, continuously, with a 3 - week (21 - day) cycle.
  The maximum treatment duration is 6 courses.

SUMMARY:
Patients with locally advanced unresectable or metastatic hepatocellular carcinoma (HCC) who progressed after prior systemic therapy (targeted ± immunotherapy) are enrolled. Primary endpoint: objective response rate (ORR). Planned enrollment: 47 subjects. Eligible patients receive adebrelimab + apatinib.

After informed consent and screening, treatment starts: Adebrelimab 1200mg IV on D1, Q3W; apatinib 250mg oral QD, continuous. 21-day cycle. Treatment continues until intolerable toxicity, consent withdrawal, RECIST v1.1-proven progression (may continue if clinically beneficial), or protocol-specified criteria (whichever first).

Safety follow-up on D1 of each cycle; imaging every 2 cycles (6-8 weeks) for efficacy. Post-treatment: continued safety and survival follow-up.

DETAILED DESCRIPTION:
In this study, patients with locally advanced unresectable or metastatic hepatocellular carcinoma who have previously received systemic therapy (targeted therapy with or without immunotherapy) and developed drug resistance and progression will be selected as the research subjects. The study takes the objective response rate (ORR) as the primary endpoint. It is planned to enroll 47 subjects. Eligible patients will receive adebrelimab in combination with apatinib for treatment.

After subjects are fully informed, sign the informed consent form, and pass the screening, they will receive the study treatment. Adebrelimab will be administered at a fixed dose of 1200 mg by intravenous infusion on D1, once every 21 days (Q3W). It will be combined with apatinib at a dose of 250 mg (0.25 g), taken orally once a day (QD), and continuously administered. A 3 - week (21 - day) period will be considered one treatment cycle. The study treatment will continue until the subject experiences intolerable toxic reactions, withdraws informed consent, disease progression confirmed by the investigator according to RECIST v1.1 (when a subject has disease progression as defined by RECIST v1.1, if the investigator assesses that the subject still has clinical benefits and can tolerate the study treatment, the subject may continue to receive the study drug; if it is considered that the subject no longer has clinical benefits, the treatment may be terminated), or other treatment termination criteria specified in the protocol, whichever occurs first.

After subjects are enrolled in the study, safety follow - up visits will be conducted on D1 of each treatment cycle. Imaging examinations will be performed once every 2 treatment cycles (6 - 8 weeks) to evaluate the efficacy. After the end of treatment, safety follow - up visits and survival follow - up will continue.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily participate in this study and sign the informed consent form;
2. Aged ≥ 18 years (calculated as of the date of signing the informed consent form), male or female;
3. Pathologically or clinically confirmed hepatocellular carcinoma (HCC);
4. Have previously received at least one or more lines of systemic therapy (targeted therapy with or without immunotherapy);
5. Barcelona Clinic Liver Cancer (BCLC) stage B or C, unsuitable for surgery or local treatment, or progressed after surgery and/or local treatment;
6. Local treatment (including but not limited to surgery, radiotherapy, hepatic artery embolization, transcatheter arterial chemoembolization [TACE], hepatic artery infusion, radiofrequency ablation, cryoablation, or percutaneous ethanol injection) must have been completed at least 4 weeks before the baseline imaging scan (palliative radiotherapy requires only 2 weeks), and toxic reactions caused by local treatment (except alopecia) must have recovered to ≤ Grade 1 according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 (NCI-CTCAE v5.0);
7. Presence of measurable lesions meeting the modified Response Evaluation Criteria in Solid Tumors (mRECIST) on baseline imaging;
8. Child-Pugh liver function class A;
9. Eastern Cooperative Oncology Group Performance Status (ECOG-PS) score of 0-1;
10. Expected survival time > 3 months;
11. Basic normal function of major organs, without severe abnormalities in blood, heart, lung, liver, kidney, bone marrow, or immunodeficiency diseases, meeting the protocol requirements:

    1. Blood routine examination: (except hemoglobin; no blood transfusion, no use of granulocyte colony-stimulating factor [G-CSF] within 14 days before screening, and no corrective treatment within 7 days) i. Hemoglobin ≥ 90 g/L; ii. Neutrophil count ≥ 1.5×10^9/L; iii. Platelet count ≥ 50×10^9/L;
    2. Biochemical examination: (no albumin transfusion within 14 days) i. Serum albumin ≥ 29 g/L; ii. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5×upper limit of normal (ULN); iii. Total bilirubin (TBIL) ≤ 1.5×ULN; iv. Creatinine (Cr) ≤ 1.5×ULN or creatinine clearance > 50 mL/min (calculated using the Cockcroft-Gault formula as follows): For males: Creatinine clearance = ((140 - age) × weight) / (72 × serum Cr) For females: Creatinine clearance = ((140 - age) × weight) / (72 × serum Cr) × 0.85 (Weight unit: kg; Serum Cr unit: mg/mL) v. Urinary protein < 2+; if urinary protein ≥ 2+, a 24-hour urinary protein quantification can be performed, and patients with 24-hour urinary protein quantification < 1.0 g are eligible for enrollment;
    3. Coagulation function: Activated partial thromboplastin time (APTT) and international normalized ratio (INR) ≤ 1.5×ULN (patients receiving stable-dose anticoagulant therapy such as low-molecular-weight heparin or warfarin with INR within the expected therapeutic range of anticoagulants can be screened);
    4. Thyroid-stimulating hormone (TSH) ≤ ULN; if abnormal, triiodothyronine (T3) and thyroxine (T4) levels should be examined, and patients with normal T3 and T4 levels are eligible;
12. Patients with active hepatitis B virus (HBV) infection who are willing to receive full-course antiviral therapy during the study (according to local standard treatment, such as entecavir) may be eligible for enrollment based on the doctor's judgment of individual patient conditions under viral load monitoring;
13. Patients with positive hepatitis C virus (HCV) ribonucleic acid (RNA) must receive antiviral therapy according to local standard treatment guidelines, and liver function elevation must be within CTCAE Grade 1;
14. Female patients of childbearing potential: Must agree to abstain from heterosexual intercourse or use reliable and effective contraception from the signing of the informed consent form until at least 120 days after the last dose of the study drug. Additionally, serum human chorionic gonadotropin (HCG) must be negative within 7 days before the start of study treatment; and must be non-lactating. A female patient is considered to have childbearing potential if she has menstruated, has not reached postmenopausal status (amenorrhea for ≥ 12 consecutive months with no other identified causes except menopause), and has not undergone sterilization (such as hysterectomy, bilateral salpingectomy, or bilateral oophorectomy);
15. Male patients whose partners are women of childbearing potential must agree to abstain from heterosexual intercourse or use reliable and effective contraception from the signing of the informed consent form until at least 120 days after the last dose of the study drug. Male subjects must also agree not to donate sperm during the same period. Male subjects whose partners are pregnant must use condoms and do not need to adopt other contraceptive methods.

Exclusion Criteria:

1. Previously received PD-L1 immunotherapy or apatinib targeted therapy;
2. No clear tumor-feeding artery identifiable by angiography;
3. Known cholangiocellular carcinoma, sarcomatoid HCC, mixed-cell carcinoma, or fibrolamellar carcinoma; having other active malignant tumors (except HCC) within 5 years or concurrently. Locally cured tumors such as basal cell carcinoma of the skin, cutaneous squamous cell carcinoma, superficial bladder cancer, carcinoma in situ of the prostate, carcinoma in situ of the cervix, and carcinoma in situ of the breast are eligible for enrollment;
4. Allergic to the investigational drugs;
5. Complicated with other malignant tumors, except for the following cases: malignant tumors treated with curative therapy, with no known active disease for ≥ 5 years before the first study intervention and low potential risk of recurrence; basal cell carcinoma of the skin, cutaneous squamous cell carcinoma, or lentigo maligna with potentially radical treatment; or carcinoma in situ with adequate treatment and no evidence of disease;
6. A history of hepatic encephalopathy;
7. Received other investigational drug treatments within 28 days or 5 half-lives (whichever is longer) before the start of study treatment;
8. Complicated with severe infection;
9. Any evidence of disease as judged by the investigator (such as severe or uncontrolled systemic diseases, including uncontrolled hypertension, active hemorrhagic diseases, active infections, active interstitial lung disease/pulmonary inflammation, severe chronic gastrointestinal diseases related to diarrhea, mental illness/social conditions) or a history of allogeneic organ transplantation that the investigator considers makes the subject unfit to participate in the study or affects compliance with the study protocol;
10. Active or previously documented autoimmune or inflammatory diseases (including inflammatory bowel diseases [e.g., colitis or Crohn's disease], diverticulitis [excluding diverticulosis], systemic lupus erythematosus, sarcoidosis syndrome, Wegener's syndrome [granulomatosis with polyangiitis], Graves' disease, rheumatoid arthritis, hypophysitis, and uveitis, etc.);
11. Known positive HIV test (positive HIV 1/2 antibodies) or active tuberculosis infection (clinical assessment may include clinical history, physical examination, and imaging findings, or tuberculosis testing according to local practices).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | up to one year
  Objective Response Rate (ORR): It refers to the percentage of subjects who achieve complete response (CR) or partial response (PR) as determined by the investigator according to RECIST v1.1, mRECIST, or imRECIST (for CR and PR under the imRECIST criteria, they can occur after radiographic disease progression).

SECONDARY OUTCOMES:
Median Progression-free survival | up to one year
  It refers to the time from the first occurrence of radiological disease progression or death (whichever comes first), as determined by the investigator in accordance with RECIST v1.1, mRECIST, or imRECIST. For radiological disease progression identified under the imRECIST criteria, if it is evaluated as response or stable disease after ≥4 weeks, this progression will not be considered a PFS event.
Time to Progression (TTP) | up to one year
  It refers to the time from the date of starting treatment to the occurrence of radiological disease progression, as determined by the investigator in accordance with RECIST v1.1, mRECIST, or imRECIST. For radiological disease progression identified under the imRECIST criteria, if it is evaluated as response or stable disease after ≥4 weeks, this progression will not be considered a TTP event.
Disease Control Rate (DCR) | up to one year
  It refers to the percentage of subjects who achieve complete response (CR), partial response (PR), or stable disease (SD) lasting for ≥8 weeks, as determined by the investigator in accordance with RECIST v1.1, mRECIST, or imRECIST (CR, PR, and SD under the imRECIST criteria can occur after radiographic disease progression).
Duration of Response (DOR) | up to one year
  It refers to the time from the first documentation of objective response (CR or PR) to the first occurrence of radiographic disease progression or death (whichever comes first), as determined by the investigator in accordance with RECIST v1.1, mRECIST, or imRECIST. For radiographic disease progression under the imRECIST criteria, if it is assessed as response or stable disease after ≥4 weeks, it will not be regarded as a progression event for DoR calculation.
Overall Survival (OS) | up to one year
  It refers to the time from randomization (or enrollment) to death from any cause.
Adverse Event (AE) | up to one year
  Adverse Event (AE) refers to all adverse medical events that occur in subjects after they receive the investigational product, which can present as symptoms, signs, diseases, or abnormal laboratory test results, but are not necessarily causally related to the investigational product. The collection of AE information starts from the time when the subject signs the informed consent form and continues until the end of the safety follow-up period (30 days after the last dose) or until the initiation of a new anti-tumor drug.
Serious Adverse Event (SAE) | up to one year
  Serious Adverse Event (SAE) refers to medical events occurring in subjects after receiving any dose of the investigational product, including those requiring hospitalization or prolongation of existing hospitalization, causing disability, impairing work capacity, endangering life, resulting in death, or leading to congenital malformations.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Science, Shenzhen Center, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No